CLINICAL TRIAL: NCT01215630
Title: Cardiovascular Fitness and Venous Function in Trained and Untrained Subjects
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2010/1512-2
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Healthy Subjects
Keywords: Veins; Exercise tests; maximal oxygen uptake; VO2max

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy subjects: Men Women Age; 18-75
  Interventions: Behavioral: Aerobic Interval Training

INTERVENTIONS:
Behavioral: Aerobic Interval Training — One interval training session

SUMMARY:
The primary aim is to study the relationship between vascular function, cardiovascular fitness and age in healthy subjects. Individuals with the highest cardiovascular fitness will have the greatest arterial inflow independent of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, 18-75 years of age

Exclusion Criteria:

* Inability to exercise due to musculoskeletal conditions
* Known ischemic cardiovascular disease
* Smoking or tobacco use
* Acute medical conditions
* Active infections
* Pharmacotherapy with known vascular effects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women, aged 18-75 yrs
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Venous Compliance | 2 weeks
  Echocardiography; Test - retest

SECONDARY OUTCOMES:
Maximal oxygen uptake | one test at baseline
  Cardiopulmonary testing

CONTACTS AND LOCATIONS:
Overall Officials: Trine Karlsen, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Leinan IM, Aamot IL, Stoylen A, Karlsen T, Wisloff U. Upper arm venous compliance and fitness in stable coronary artery disease patients and healthy controls. Clin Physiol Funct Imaging. 2017 Sep;37(5):498-506. doi: 10.1111/cpf.12324. Epub 2015 Dec 15. PMID 26667796
- [Result] Leinan IM, Grønnevik Ø, Støylen A, Wisløff U, Karlsen T. A cross sectional study of arm venous compliance in fit healthy subjects. Journal of Cardiovascular Research 1(2). http://www.vipoa.org/journals/pdf/5947267721.pdf